CLINICAL TRIAL: NCT00331448
Title: Fat Redistribution and Metabolic Change in HIV Infection (FRAM)
Brief Title: Observational Study of Changes in Fat Distribution and Blood Metabolites in HIV Infected Adults
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute on Drug Abuse (NIDA) (NIH); NIH Office of AIDS Research (OAR) (NIH)
Other Study IDs: DK-57508 / HL-74814; DK-57508; HL-74814
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-05

CONDITIONS: HIV Infections; Lipodystrophy; Diabetes; Hyperlipidemia; Atherosclerosis
Keywords: Treatment Experienced; Lipoatrophy; Lipohypertrophy; Glucose; Cholesterol; Triglycerides; MRI; DXA; Carotid IMT; LDL; HDL
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Diabetes Mellitus; Hyperlipidemias; Atherosclerosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to collect data on the body's breakdown of sugar and fat in HIV infected adults. Data from this study will make clearer the roles of HIV infection and anti-HIV drugs in the development of diabetes, heart disease, and fat redistribution in HIV infected adults.

DETAILED DESCRIPTION:
Changes in the amount of fat and how that fat was distributed were reported after the introduction of antiretroviral therapy (ART) for HIV infected patients. Increases in diabetes, heart disease, and blood levels of glucose and fats have also been reported. However, the cause for these changes is still unclear, in part because clinical measures have not been consistent between different trials. The contribution of age, duration of HIV infection, duration and types of ART, and body weight on metabolic changes need to be defined, and the relationship between metabolic disturbances and body composition changes has also not been established. The purpose of this study is to examine HIV infected adults and use objective measurements of fat to determine metabolic changes in this population, their causes, and possible associations with other observed changes. Data from this study will help guide future treatment plans for HIV infected people to help prevent or lessen the risk for diabetes and cardiovascular disease.

There are 2 parts to this study. Part 1 will examine fat redistribution; there will be 2 groups in Part 1. Group 1 participants will be HIV infected adults recruited from specific HIV clinics. Group 2 participants will be HIV uninfected adults currently enrolled in the Coronary Artery Risk Development in Young Adults (CARDIA) study. Participants will undergo hands-over-head-to-toe wide-slice magnetic resonance imaging (MRI) and dual energy x-ray absorptiometry (DEXA). Imaging measurements will be compared to anthropometric measurements to determine whether anthropometric measurements can accurately quantify fat redistribution. Participants will be asked to self-report fat distribution abnormalities, and this self-reporting will be evaluated for accuracy as compared to the quantitative measures of regional fat distribution. Blood collection will also occur to determine the possible association of body composition changes with the types of ART a participant may have taken or currently be taking.

Part 2 of this study will examine cardiovascular disease and factors for its development; there will be 2 groups in Part 2. Group 1 participants will be HIV infected adults recruited from specific HIV clinics. Group 2 participants will be HIV uninfected adults currently enrolled in the CARDIA study. All participants will be assessed for blood pressure, family history, lifestyle habits, and regional fat volumes by MRI and DEXA. Blood collection will occur to test for glucose and lipids (traditional metabolic risk factors) and C-reactive protein (CRP) and cytokines (novel inflammatory risk factors). Participants will also undergo a carotid intimal medial thickness (IMT) measurement by ultrasound to determine the prevalence of atherosclerosis in this population and associated contributing factors.

For Part 2, there will be a minimum of 2 visits. At both visits, fasting blood collection will occur. A physical exam and self-reporting of lifestyle habits, and completion of questionnaires about smoking, alcohol use, and medical and family history will occur at the first visit.

ELIGIBILITY:
Inclusion Criteria for Group 1 in Parts 1 and 2:

* HIV infected
* Recruited from an HIV clinic participating in this study

Inclusion Criteria for Group 2 in Parts 1 and 2:

* HIV uninfected
* Participating in the CARDIA study

Exclusion Criteria:

* Inability to undergo DEXA and MRI studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1483
Dates: Start 2000-06; Study Completion 2007-07

CONTACTS AND LOCATIONS:
Overall Officials: Carl Grunfeld, MD, PhD, Principal Investigator — Northern California Institute for Research and Education, University of California, San Francisco, Veterans Affairs Medical Center

REFERENCES:
- [Background] Safrin S, Grunfeld C. Fat distribution and metabolic changes in patients with HIV infection. AIDS. 1999 Dec 24;13(18):2493-505. doi: 10.1097/00002030-199912240-00002. No abstract available. PMID 10630518
- [Result] Bacchetti P, Gripshover B, Grunfeld C, Heymsfield S, McCreath H, Osmond D, Saag M, Scherzer R, Shlipak M, Tien P; Study of Fat Redistribution and Metabolic Change in HIV Infection (FRAM). Fat distribution in men with HIV infection. J Acquir Immune Defic Syndr. 2005 Oct 1;40(2):121-31. doi: 10.1097/01.qai.0000182230.47819.aa. PMID 16186728
- [Result] Study of Fat Redistribution and Metabolic Change in HIV Infection (FRAM). Fat distribution in women with HIV infection. J Acquir Immune Defic Syndr. 2006 Aug 15;42(5):562-71. doi: 10.1097/01.qai.0000229996.75116.da. PMID 16837863
- [Derived] Scherzer R, Heymsfield SB, Rimland D, Powderly WG, Tien PC, Bacchetti P, Shlipak MG, Grunfeld C; Study of Fat Redistribution, Metabolic Change in HIV Infection (FRAM). Association of serum albumin and aspartate transaminase with 5-year all-cause mortality in HIV/hepatitis C virus coinfection and HIV monoinfection. AIDS. 2017 Jan 2;31(1):71-79. doi: 10.1097/QAD.0000000000001278. PMID 27677166
- [Derived] Wheeler AL, Scherzer R, Lee D, Delaney JA, Bacchetti P, Shlipak MG, Sidney S, Grunfeld C, Tien PC; Study of Fat Redistribution and Metabolic Change in HIV Infection (FRAM). HIV/hepatitis C virus coinfection ameliorates the atherogenic lipoprotein abnormalities of HIV infection. AIDS. 2014 Jan 2;28(1):49-58. doi: 10.1097/QAD.0000000000000026. PMID 24136113
- [Derived] Kosmiski LA, Scherzer R, Heymsfield SB, Rimland D, Simberkoff MS, Sidney S, Shlipak MG, Bacchetti P, Biggs ML, Grunfeld C; Study of Fat Redistribution and Metabolic Change in HIV Infection (FRAM). Association of increased upper trunk and decreased leg fat with 2-h glucose in control and HIV-infected persons. Diabetes Care. 2011 Nov;34(11):2448-53. doi: 10.2337/dc11-0616. Epub 2011 Sep 16. PMID 21926283
- [Derived] Scherzer R, Heymsfield SB, Lee D, Powderly WG, Tien PC, Bacchetti P, Shlipak MG, Grunfeld C; Study of Fat Redistribution and Metabolic Change in HIV Infection (FRAM). Decreased limb muscle and increased central adiposity are associated with 5-year all-cause mortality in HIV infection. AIDS. 2011 Jul 17;25(11):1405-14. doi: 10.1097/QAD.0b013e32834884e6. PMID 21572308
- [Derived] Jotwani V, Scherzer R, Choi A, Szczech L, Polak JF, Kronmal RA, Grunfeld C, Shlipak M. Reduced kidney function and preclinical atherosclerosis in HIV-infected individuals: the study of fat redistribution and metabolic change in HIV infection (FRAM). Am J Nephrol. 2011;33(5):453-60. doi: 10.1159/000327606. Epub 2011 Apr 21. PMID 21508633
- [Derived] Delaney JA, Scherzer R, Biggs ML, Shliplak MG, Polak JF, Currier JS, Kronmal RA, Wanke C, Bacchetti P, O'leary D, Tien PC, Grunfeld C. Associations of antiretroviral drug use and HIV-specific risk factors with carotid intima-media thickness. AIDS. 2010 Sep 10;24(14):2201-9. doi: 10.1097/QAD.0b013e32833d2132. PMID 20671544
- [Derived] Tien PC, Choi AI, Zolopa AR, Benson C, Tracy R, Scherzer R, Bacchetti P, Shlipak M, Grunfeld C. Inflammation and mortality in HIV-infected adults: analysis of the FRAM study cohort. J Acquir Immune Defic Syndr. 2010 Nov;55(3):316-22. doi: 10.1097/QAI.0b013e3181e66216. PMID 20581689
- [Derived] Scherzer R, Shen W, Heymsfield SB, Lewis CE, Kotler DP, Punyanitya M, Bacchetti P, Shlipak MG, Grunfeld C; Study of Fat Redistribution and Metabolic Change in HIV Infection (FRAM). Intermuscular adipose tissue and metabolic associations in HIV infection. Obesity (Silver Spring). 2011 Feb;19(2):283-91. doi: 10.1038/oby.2010.115. Epub 2010 Jun 10. PMID 20539305
- [Derived] Cockerham L, Scherzer R, Zolopa A, Rimland D, Lewis CE, Bacchetti P, Grunfeld C, Shlipak M, Tien PC. Association of HIV infection, demographic and cardiovascular risk factors with all-cause mortality in the recent HAART era. J Acquir Immune Defic Syndr. 2010 Jan;53(1):102-6. doi: 10.1097/QAI.0b013e3181b79d22. PMID 19738484
- [Derived] Grunfeld C, Delaney JA, Wanke C, Currier JS, Scherzer R, Biggs ML, Tien PC, Shlipak MG, Sidney S, Polak JF, O'Leary D, Bacchetti P, Kronmal RA. Preclinical atherosclerosis due to HIV infection: carotid intima-medial thickness measurements from the FRAM study. AIDS. 2009 Sep 10;23(14):1841-9. doi: 10.1097/QAD.0b013e32832d3b85. PMID 19455012
- [Derived] Grunfeld C, Rimland D, Gibert CL, Powderly WG, Sidney S, Shlipak MG, Bacchetti P, Scherzer R, Haffner S, Heymsfield SB. Association of upper trunk and visceral adipose tissue volume with insulin resistance in control and HIV-infected subjects in the FRAM study. J Acquir Immune Defic Syndr. 2007 Nov 1;46(3):283-90. doi: 10.1097/qai.0b013e31814b94e2. PMID 18167644